CLINICAL TRIAL: NCT03070795
Title: Outcomes of Early Versus Delayed Oral Feeding After Elective Cesarean Section in a Teaching Hospital in Ghana.
Brief Title: Outcomes of Early Versus Delayed Oral Feeding After Cesarean Section in Korle-bu Teaching Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ghana Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KBTH - IRB /00065/2016
Record Dates: First submitted 2017-02-17; First posted 2017-03-06 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Cesarean Section Complications
Keywords: post-operative ileus; early feeding; delayed feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early feeding (Experimental): patients undergoing elective cesarean section will be allowed to feed (sips) four hours after cesarean section.
  Interventions: Procedure: early feeding
- delayed feeding (Active Comparator): patients undergoing elective cesarean section will be allowed to feed on post operation day 1 (12 hours post op).
  Interventions: Procedure: delayed feeding

INTERVENTIONS:
Procedure: early feeding — start oral sips four hours after cesarean section
  Arms: early feeding
Procedure: delayed feeding — start oral feeding on post operation day 1 (>12hours) after surgery
  Arms: delayed feeding

SUMMARY:
study compares the outcomes of feeding mothers early (4 hours ) after cesarean section compared to delayed feeding (on post operation day 1) in terms of gastrointestinal function and maternal satisfaction with the feeding schedule.

DETAILED DESCRIPTION:
patients who are scheduled to undergo elective cesarean section are randomised to two groups, one group will be allowed to feed 4 hours after cesarean section while the other group will be fed traditionally by feeding on the first post op day. gastrointestinal signs and symptoms will be measured such as post operative ileus, vomiting, nausea, abdminal distension. other parameters to be measured include time to ambulate out of bed after surgery, time to start breastfeeding after surgery. satisfaction with both feeding regimes will be assessed after surgery and the incedence of wound infecion will be compared between the two groups after two weeks durung the post natal review.

ELIGIBILITY:
Inclusion Criteria:

Uncomplicated elective Cesarean sections performed under regional anaesthesia without extensive intra operative bowel adhesions.

Women who give consent to participate in the study.

Exclusion Criteria:

* Elective Cesarean sections complicated by severe haemorrhage, bowel injury requiring bowel manipulation, repair, resection and anastomosis or colostomy.

Women who require a Cesarean hysterectomy. Women who require a Post-partum hysterectomy. Mothers with severe pre-eclampsia. Mothers with sickle cell disease. Mothers with pregestational or gestational diabetes. Mothers who have been scheduled for Cesarean section and require general anaesthesia.

Women who have had a previous laparotomy other than a Cesarean section.

Max Age: 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-06-20 (Estimated); Study Completion 2017-08-20 (Estimated)

PRIMARY OUTCOMES:
post-operative ileus | within 3 days after surgery
  onset of vomiting >4 times per day

SECONDARY OUTCOMES:
Crampy abdominal pain | within 3 days after surgery
  abdominal pain after feeding following cesarean section
Time of initiation of breastfeeding post operatively | within 3 days after surgery
  time it takes to start breastfeeding after cesrean section
Woman's satisfaction | within 3 days after surgery
  measure level of satisfaction with feeding regime using an assessment scoring tool. this is in the form of a questionair adminstered to the client by the investigator.
Time of ambulation out of bed after surgery | within 3 days after surgery
  time it takes for the mother to get out of bed and sit up or mobilize
Incedence of a wound infection | within 2 weeks of surgery
  measure of the presence of wound infection in both arms on day of discharge and 2 weeks post discharge

CONTACTS AND LOCATIONS:
Overall Officials: kojo apea-kubi, Principal Investigator — Korle Bu Teaching Hospital; isaac abiaw, Principal Investigator — Korle Bu Teaching Hospital
Locations (1):
- Korle-Bu Teaching Hospital, Accra, Greater Accra Region, Ghana

IPD SHARING:
Plan to Share IPD: Undecided